CLINICAL TRIAL: NCT03671382
Title: Training Oncologists and Empowering Patients in Affective Communication During Medical Consultations in Singapore (TEAMS) - A Pilot Study
Brief Title: Communication During Medical Consultations in Singapore -Pilot
Acronym: TEAMS-pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Chetna Malhotra, Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCPC-IN
Record Dates: First submitted 2018-09-02; First posted 2018-09-14 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Communication Research
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Communication Training Program and Patient Prompt Sheet
  Interventions: Behavioral: Communication Training Program and Patient Prompt Sheet
- Control Arm (No Intervention): Oncologists will not receive the communication skills training program and their patients will not receive the Patient Prompt Sheet

INTERVENTIONS:
Behavioral: Communication Training Program and Patient Prompt Sheet — The intervention being delivered is a two-component intervent. First component is the Oncologist Communication Skills Training Program. This is an e-learning module teaching oncologists to recognize and respond to patient/caregiver distress, provide information including prognosis and discuss goals of care. The second component is a patient prompt sheet which will be administered to three patients of intervention arm oncologists in the waiting area at least 30 minutes before their consultation. The sheet includes structured questions for patients to ask the oncologist about diagnosis and prognosis and will prompt patients to label and express their emotions in a direct manner.
  Arms: Intervention Arm

SUMMARY:
Despite advanced cancer patients and their caregivers frequently experiencing psychological distress and wanting to know about their prognosis, oncologists rarely respond with empathy and provide adequate information regarding patient prognosis. We aim to address the communication gap during consultations by developing an Oncologist E-Learning Communications Skills Training Program guiding physicians on how to recognize and respond to patient/caregiver distress and to disclose prognosis; and a Patient Prompt Sheet to encourage discussions of psychological distress and prognosis. We will assess the feasibility of delivering this two-component intervention program within a cancer center in Singapore through a 2-arm randomized controlled trial in which 8 oncologists will be randomly assigned to Control Arm (n=4) and Intervention Arm (n=4). Oncologists in the intervention arm will receive the E-Learning Program. Their patients will also receive the Patient Prompt Sheet before their consultation with oncologist. After completion of oncologist intervention we will audio-record and survey 3 patients with Stage IV cancer and their caregivers per oncologist before and after their consultations. If the study is shown to be feasible and acceptable, then its effectiveness will be assessed in a larger trial.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for oncologists are

1. All consultants and senior residents/registrars in the Departments of Medical Oncology at National Cancer Centre, Singapore
2. Able to allow audio-recording during consultation

The inclusion criteria for patients are

1. Age ≥ 21 years old
2. Patients who are consulting an oncologist who is participating in the study
3. Patients who are Singaporeans or Singapore Permanent Residents
4. Diagnosis of stage IV cancer (with metastasis to visceral organs)
5. Able to allow audio-recording during consultation

Exclusion Criteria:

The exclusion criteria for oncologists are

a. Rejecting audio-recording during consultation

The exclusion criteria for patients are

1. Age ≤ 21 years old
2. Patients who are not Singaporeans or Singapore Permanent Residents
3. Rejecting audio-recording during consultation
4. Patients with psychiatric or cognitive disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Assess feasibility and acceptability of intervention | up to 3 months
  Measured by proportion of intervention arm oncologists completing their intervention

SECONDARY OUTCOMES:
Assess increase in number of empathic statements by oncologists | within 5 months
  Measured by coding audio-recorded consultations post-intervention
Assess increase in number of questions related to their prognosis asked by patients | within 5 months
  Measured by coding audio-recorded consultations post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chetna Malhotra, MD, MPH, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No